CLINICAL TRIAL: NCT00472056
Title: Randomized Trial Using Standard Dose Versus High Dose Rituximab in Addition to Autologous Transplantation With BEAM for Patients With Diffuse Large B Cell Lymphomas
Brief Title: Rituximab in Addition to Autologous Transplantation With BEAM for Patients With Lymphoid Malignancies
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2004-0271
Record Dates: First submitted 2007-05-09; First posted 2007-05-11 (Estimated); Results first posted 2012-02-13 (Estimated); Last update posted 2016-03-15 (Estimated); Status verified 2012-06

CONDITIONS: Lymphoma
Keywords: Non-Hodgkin's Lymphoma; Lymphoid Malignancies; Lymphoma; BEAM Chemotherapy; Carmustine; BCNU; BiCNU; Etoposide; VePesid; Cytarabine; Cytosar; DepoCyt; Cytosine arabinosine hydrochloride; Ara-C; Melphalan; Rituximab; Rituxan
MeSH Terms: conditions — Lymphoma; Lymphoma, Non-Hodgkin | interventions — Carmustine; Etoposide; Cytarabine; Melphalan; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BEAM + Standard Rituximab (Experimental): Arm 1 BEAM Chemotherapy (Carmustine, Etoposide, Cytarabine, Melphalan) + Standard Rituximab with Standard Rituximab for Cohort 1 or 2
  Cohort 1 for 65 years of age or younger BEAM: Carmustine 300 mg/m2 intravenous (IV) over 1 hour on day -6, cytarabine 200 mg/m2 IV twice a day on days -5 through -2 (total 8 doses), etoposide 200 mg/m2 IV twice a day on days -5 through -2 (total 8 doses), and melphalan 140 mg/m2 IV on day -1.
  Cohort 2 for older than 65 years of age BEAM: Carmustine 300 mg/m2 IV over 1 hour on day -6, cytarabine 100 mg/m2 IV twice a day on days -5 through -2 (total 8 doses), etoposide 100 mg/m2 IV twice a day on days -5 through -2 (total 8 doses), and melphalan 140 mg/m2 IV on day -1.
  Standard Rituximab: 375 mg/m^2 IV Days +1, +8 after Stem Cell Infusion on Day 0.
  Interventions: Drug: Carmustine; Drug: Etoposide; Drug: Cytarabine; Drug: Melphalan; Drug: Rituximab
- BEAM + High Rituximab (Experimental): BEAM Chemotherapy (Carmustine, Etoposide, Cytarabine, Melphalan) + High Dose Rituximab
  Cohort 1 for 65 years of age or younger BEAM: Carmustine 300 mg/m2 intravenous (IV) over 1 hour on day -6, cytarabine 200 mg/m2 IV twice a day on days -5 through -2 (total 8 doses), etoposide 200 mg/m2 IV twice a day on days -5 through -2 (total 8 doses), and melphalan 140 mg/m2 IV on day -1.
  Cohort 2 for older than 65 years of age BEAM: Carmustine 300 mg/m2 IV over 1 hour on day -6, cytarabine 100 mg/m2 IV twice a day on days -5 through -2 (total 8 doses), etoposide 100 mg/m2 IV twice a day on days -5 through -2 (total 8 doses), and melphalan 140 mg/m2 IV on day -1.
  High Dose Rituximab: 1000 mg/m^2 IV Days +1, +8 after Stem Cell Infusion on Day 0
  Interventions: Drug: Carmustine; Drug: Etoposide; Drug: Cytarabine; Drug: Melphalan; Drug: Rituximab

INTERVENTIONS:
Drug: Carmustine — 300 mg/m^2 IV for 1 Day
  Other Names: BCNU; BiCNU
Drug: Etoposide — Arm 1 = 200 mg/m^2 IV Every 12 Hours x 4 Days; Arm 2 = 100 mg/m^2 IV Every 12 Hours x 4 Days
  Other Names: VePesid
Drug: Cytarabine — Arm 1 = 200 mg/m^2 IV Every 12 Hours x 4 Days; Arm 2 = 100 mg/m^2 IV Every 12 Hours x 4 Days
  Other Names: Ara-C; Cytosar; DepoCyt; Cytosine arabinosine hydrochloride
Drug: Melphalan — 140 mg/m^2 IV x 1 Day
Drug: Rituximab — Cohort 1, High-Dose Rituximab = 1000 mg/m^2 IV On Days +1 and +8 After Stem Cell Infusion; Cohort 2, Standard Dose Rituximab = 375 mg/m^2 IV On Days +1 and +8 After Stem Cell Infusion.
  Other Names: Rituxan

SUMMARY:
Cohort 1: Patients who are less than or equal to 65 years of age.

1. To determine the disease-free survival (DFS) in the 2 arms (standard dose versus high dose rituximab)

Cohort 2: Patients who are older than 65 years of age

1. To determine the disease-free survival (DFS) in the 2 arms (standard dose versus high dose rituximab)
2. To determine the treatment related mortality (TRM)

DETAILED DESCRIPTION:
Carmustine, cytarabine, etoposide, melphalan, and rituximab are all standard chemotherapy drugs.

If you are found to be eligible to take part in this study, you will be randomly assigned (as in the toss of a coin) to one of two treatment groups. Participants in one group will receive high dose rituximab with transplantation and high dose chemotherapy. Participants in the other group will receive standard dose rituximab with transplantation and high dose chemotherapy. The first 10 patients enrolled on this study will have an equal chance of being assigned to either group. After the first 10 participants are enrolled, the remaining participants will have a higher chance of being assigned to the group that has proven to be more effective.

All participants will have a plastic tube (catheter) inserted under their collarbone. This catheter will be left in place for the entire treatment period. The catheter will be used to deliver most of the drugs and for the collection and transfusion of the stem cells. When possible, all drugs that need to be given by vein will be given using the catheter.

Stem cell collection is done on a separate study and patients will take part in this study only after the stem cell collection is complete. You should have an adequate number of stem cells collected and stored before you can be eligible for high-dose chemotherapy and transplantation.

All treatment will be given at M. D. Anderson. You will be admitted to the hospital to receive high dose chemotherapy and will stay in the hospital for 3-4 weeks. You will be given carmustine by vein over 1 hour on Day 1. On Days 2 - 5, you will be given cytarabine by vein over 1 hour and etoposide by vein over 3 hours. This will be repeated every 12 hours on Days 2-5. On Day 6, you will be given melphalan by vein over 30 minutes. On Day 7, the stem cells that were collected earlier will be given back to you ("transplanted") through the catheter over 30-45 minutes.

You will also receive either high dose or standard dose rituximab by vein over 4-6 hours one day after the transplant (Day 1) and then again 1 week later (Day 8).

You will receive G-CSF injections staring at Day 1 (one day after transplant or stem cell infusion). These will continue our cell count reaches the appropriate level for at least 3 days in a row. Blood tests (2 teaspoons) will be done every day while you are in the hospital to track the effects of the transplant.

You will be asked to return to M. D. Anderson at 3 months and 6 months after transplantation, then every 6 months for 3 years, and then once a year up to 5 years from the transplant date. At each visit you will get blood work (1-2 tablespoons), CT scans, and other tests like bone marrow (if needed) to determine the status of your lymphoma.

This is an investigational study. All of the drugs used in this study are FDA approved and are commercially available. Up to 100 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically proven diffuse large B-cell (CD20 positive) or transformed follicular non-Hodgkin's lymphomas, that have relapsed after conventional chemotherapy and are not eligible for protocols of higher priority
2. Patients must have chemosensitive disease to salvage chemotherapy and less than 5% bone marrow involvement with lymphoma by gross pathologic examination
3. Age less than or equal to 80 years. There is no lower age limit for this study.
4. Zubrod performance status of less than 2
5. Negative pregnancy test in patients with child bearing potential
6. Must be willing to sign informed consent
7. Should be seronegative for HIV, hepatitis B surface antigen, hepatitis C antibody.

Exclusion Criteria:

1. Patients with known active CNS disease are excluded. Patients with prior history of CNS disease should have a negative MRI of the brain (and/or spine if indicated) and negative CSF cytology within 4 weeks of enrollment into the study.
2. Less than 3 weeks from last cytotoxic chemotherapy
3. Serum bilirubin > 1.5 mg/dl
4. Serum transaminases > 2X/ULN
5. Serum creatinine > 1.6 mg/dl
6. Failure to collect more than 3 x 1,000,000 CD34+ stem cells/kg body weight
7. Left ventricular ejection fraction of < 40%, unless cleared by cardiology
8. Corrected DLCO of < 50%
9. Patients who are on anticoagulants or antiplatelet agents.

Max Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2005-03; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chitra M. Hosing, MD, Principal Investigator — UT MD Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: March 03, 2005 to June 19, 2009. All recruitment done at UT MD Anderson Cancer Center.
Groups:
- Cohort 1 65 Years of Age or Less With Arm 2; Cohort 2 Patients Who Are Older Than 65 Years of Age Arm 2: Arm 2: BEAM Chemotherapy (Carmustine, Etoposide, Cytarabine, Melphalan) + High Dose Rituximab
- Cohort 2 Patients Who Are Older Than 65 Years of Age Arm 1; Cohort 1 65 Years of Age or Less With Arm 1: Arm 1: BEAM Chemotherapy (Carmustine, Etoposide, Cytarabine, Melphalan) + Standard Dose Rituximab
Period: Overall Study
Arm/Group | Cohort 1 65 Years of Age or Less With Arm 2 | Cohort 2 Patients Who Are Older Than 65 Years of Age Arm 1 | Cohort 1 65 Years of Age or Less With Arm 1 | Cohort 2 Patients Who Are Older Than 65 Years of Age Arm 2
Started | 25 | 19 | 32 | 17
Completed | 25 | 19 | 32 | 17
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 65 Years of Age or Less With Arm 2 | Cohort 2 Patients Who Are Older Than 65 Years of Age Arm 1 | Cohort 1 65 Years of Age or Less With Arm 1 | Cohort 2 Patients Who Are Older Than 65 Years of Age Arm 2 | Total
Number analyzed (Participants) | 25 | 19 | 32 | 17 | 93
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 1 | 0 | 1
  Between 18 and 65 years | 25 | 0 | 31 | 0 | 56
  >=65 years | 0 | 19 | 0 | 17 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.6 (7.58288) | 70.2 (3.50522) | 53.3 (11.93155) | 69.8 (3.43211) | 61 (11.17466)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 2 | 11 | 4 | 27
  Male | 15 | 17 | 21 | 13 | 66
Region of Enrollment [Number; unit: participants]
  United States | 25 | 19 | 32 | 17 | 93

OUTCOME MEASURES:

1. Primary Outcome: Disease-free Survival (DFS)
Description: DFS defined as time from transplantation to disease relapse, disease progression, death during remission, or last follow-up. Evaluation at 3 months and 6 months after transplantation, then every 6 months for 3 years, and then once a year up to 5 years from the transplant date.
Time Frame: Up to 5 years from transplant date.
Population: Analysis was per protocol.
Measure: Mean (Full Range); unit: months
Groups:
- Standard Dose Rituximab: Standard dose arm: Rituximab 375 mg/m^2 intravenous on days +1 and +8 after stem cell infusion.
- High Dose Rituximab: High dose arm: Rituximab 1000mg/m^2 intravenous on days +1 and +8 after stem cell infusion
Arm/Group | Standard Dose Rituximab | High Dose Rituximab
Number analyzed (Participants) | 51 | 42
months | 11.33 [1.81 to 39.29] | 9.635 [1.77 to 31.45]

ADVERSE EVENTS:
Time Frame: 4 Years, 5 Months
Arm/Group | Cohort 1 65 Years of Age or Less With Arm 2 | Cohort 2 Patients Who Are Older Than 65 Years of Age Arm 1 | Cohort 1 65 Years of Age or Less With Arm 1 | Cohort 2 Patients Who Are Older Than 65 Years of Age Arm 2
Serious Adverse Events (participants affected / at risk) | 14/25 | 9/19 | 9/32 | 8/17
Other Adverse Events (participants affected / at risk) | 24/25 | 18/19 | 31/32 | 16/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 65 Years of Age or Less With Arm 2 (N=25) | Cohort 2 Patients Who Are Older Than 65 Years of Age Arm 1 (N=19) | Cohort 1 65 Years of Age or Less With Arm 1 (N=32) | Cohort 2 Patients Who Are Older Than 65 Years of Age Arm 2 (N=17)
Mucositis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutropenic fever (Infections and infestations) | 9 (9) | 6 (7) | 8 (8) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0) | 1 (1)
Renal Insufficiency (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 4 (6) | 2 (2) | 3 (6) | 3 (5)
Hyperbilirubinemia (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Transaminitis (Hepatobiliary disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Low Platelets (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Failure to Thrive (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 65 Years of Age or Less With Arm 2 (N=25) | Cohort 2 Patients Who Are Older Than 65 Years of Age Arm 1 (N=19) | Cohort 1 65 Years of Age or Less With Arm 1 (N=32) | Cohort 2 Patients Who Are Older Than 65 Years of Age Arm 2 (N=17)
Nausea (Gastrointestinal disorders) | 15 (15) | 12 (12) | 25 (25) | 12 (12)
Diarrhea (Gastrointestinal disorders) | 18 (18) | 8 (8) | 21 (21) | 9 (9)
Mucositis (Gastrointestinal disorders) | 19 (19) | 6 (6) | 28 (28) | 11 (11)
Renal Insufficiency (Renal and urinary disorders) | 0 (0) | 3 (3) | 2 (2) | 1 (1)
Transaminitis (Hepatobiliary disorders) | 1 (1) | 2 (3) | 5 (6) | 1 (1)
Hyperbilirubinemia (Hepatobiliary disorders) | 1 (1) | 4 (4) | 6 (6) | 7 (7)
Fever (Infections and infestations) | 2 (3) | 0 (0) | 1 (1) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 5 (5) | 1 (1) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes